CLINICAL TRIAL: NCT00863109
Title: Evaluation of the Health-Related Quality of Life During Combined Treatment of Chronic Hepatitis Due to Hepatitis C Virus Under Habitual Clinical Practise Conditions.
Brief Title: Quality of Life During Treatment of Chronic Hepatitis C (P05278/MK-4031-336)
Acronym: VIDA
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05278; MK-4031-336 (Other: Merck)
Record Dates: First submitted 2009-03-12; First posted 2009-03-17 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic; Genotype 1; HCV-1
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEG + RBV (Standard Clinical Practice): Participants receive peginterferon alfa-2b (PEG) and ribavirin (RBV) in combination therapy for 48 weeks according to standard clinical practice followed by 24 weeks of observation.
  Interventions: Biological: Peginterferon alfa-2b (PEG); Drug: Ribavirin (RBV)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (PEG) — Pegylated interferon alfa-2b was administered in accordance with the dosage and pattern prescribed by each participant's physician (standard clinical practice).
  Other Names: PegIntron; SCH 054031
Drug: Ribavirin (RBV) — Ribavirin was administered in accordance with the dosage and pattern prescribed by each participant's physician (standard clinical practice).
  Other Names: Rebetol; SCH 18908

SUMMARY:
The primary objective of this study is to evaluate the impact of chronic hepatitis C (CHC), and the treatment thereof with peginterferon alpha-2b (PEG) and ribavirin (RBV) according to standard clinical practice, on the health-related quality of life (HRQL) of a cohort of participants throughout 72 weeks of follow-up. HRQL was assessed using the 36-Item Short-Form Health Survey (SF-36) and the Chronic Liver Disease Questionnaire-Hepatitis C Virus (CLDQ-HCV).

DETAILED DESCRIPTION:
As widely shown in previous reports Hepatitis C Virus (HCV) patients commonly experience fatigue, anxiety, and depression. These symptoms negatively affect patients' functional health, ability to work, self-perceived health, HRQL and well-being. Psychosocial issues and reduced HRQL are frequently experienced by HCV patients. HCV patients have more HRQL impairment than the general population. There is some evidence that HCV patients who experience greater fatigue, greater psychiatric symptoms, and poorer HRQL are more likely to discontinue treatment prematurely, with a negative impact on virological response. In addition to well-known side effects of interferon, one important determinant of HRQL during anti-viral therapy for HCV is development of RBV-induced anemia. Treatment of anemia improves HRQL, potentially impacting adherence to antiviral regimen and improving virologic response. These issues emphasize the importance of investigating the physical and psychosocial experiences and HRQL of HCV patients.

The sample size of the study must allow evaluating HRQL of HCV patients based on the SF-36 before PEG treatment and at each of the following study visits.

To be able to detect differences of or over 4.2 points in the vitality dimension between the basal visit and following visits, estimating a standard deviation of 22 points, a statistical power of 80%, and a level of significance of 0.05, 216 patients will be needed. Considering a loss of follow up of 15%, a total of 238 patients are planned for this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with chronic hepatitis C (CHC)
* Participants with HCV genotype 1
* Participants who, at the time of the study, are referred to the Hospital Pharmacy Service to begin treatment with PEG and RBV for 48 weeks
* Available to understand and to give Informed Consent

Exclusion Criteria:

- Participants co-infected with Human Immunodeficiency Virus (HIV) or Hepatitis B Virus (HBV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Chronic Hepatitis C, Genotype 1, no other co-infection and compensated liver disease who receive PEG and RBV in combination therapy according to standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05278&kw=P05278&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 133 participants who enrolled on study, 3 participants failed screening and 130 were evaluable for this study.
Period: Treatment Period
Arm/Group | PEG + RBV (Standard Clinical Practice)
Started | 130
Completed | 53
Not Completed | 77
Period: Follow-up Period
Arm/Group | PEG + RBV (Standard Clinical Practice)
Started | 59 (Follow-up performed on 53 who completed Treatment Period plus 6 who discontinued treatment)
Completed | 48
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: Of 133 enrolled participants, Baseline Characteristics were reported for 130 evaluable participants. 3 enrolled participants who failed screening did not have Baseline Characteristics reported.
Groups:
- PEG + RBV (Standard Clinical Practice): Participants receive PEG and RBV in combination therapy for 48 weeks according to standard clinical practice followed by 24 weeks of observation.
Arm/Group | PEG + RBV (Standard Clinical Practice)
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 67

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) to Week 72 (WK72) in 36-Item Short-Form Health Survey (SF-36) Scores
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: physical component summary (PCS) and mental component summary (MCS). The SF-36 consists of 8 subscales. The PCS is represented by 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL. PCS and MCS scores are constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score; higher scores indicate better health status.
Time Frame: Baseline, Week 72
Population: All Evaluable Participants (participants who had met the evaluation and eligibility criteria and were included in the study) who had SF-36 data available at baseline and Week 72.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEG + RBV (Standard Clinical Practice)
Number analyzed (Participants) | 126
score on a scale
  Physical Function-BL (n=123) | 87.27 (20.67)
  Physical Function-WK72 (n=45) | 87.33 (16.08)
  Physical Function Change from BL (n=45) | -1.56 (16.30)
  Physical Role-BL (n=123) | 81.71 (36.08)
  Physical Role-WK72 (n=45) | 86.67 (29.48)
  Physical Role Change from BL (n=45) | -0.56 (35.15)
  Pain-BL (n=126) | 77.88 (23.96)
  Pain-WK72 (n=46) | 82.35 (21.41)
  Pain Change from BL (n=46) | -2.22 (19.09)
  General Health-BL (n=122) | 62.22 (18.83)
  General Health-WK72 (n=46) | 66.24 (23.24)
  General Health Change from BL (n=46) | 1.86 (19.52)
  Vitality-BL (n=121) | 67.20 (22.23)
  Vitality-WK72 (n=45) | 68.33 (19.80)
  Vitality Change from BL (n=45) | -4.30 (21.51)
  Social Function-BL (n=126) | 81.55 (23.75)
  Social Function-WK72 (n=46) | 86.96 (19.71)
  Social Function Change from BL (n=46) | 2.17 (22.56)
  Emotional Role-BL (n=123) | 79.95 (37.63)
  Emotional Role-WK72 (n=45) | 87.41 (30.39)
  Emotional Role Change from BL (n=45) | 1.48 (39.54)
  Mental Health-BL (n=121) | 71.55 (19.70)
  Mental Health-WK72 (n=45) | 74.76 (20.29)
  Mental Health Change from BL (n=45) | 1.16 (19.38)
  PCS-BL (n=121) | 50.40 (7.90)
  PCS-WK72 (n=45) | 50.73 (6.82)
  PCS Change from BL (n=45) | -0.90 (6.38)
  MCS-BL (n=121) | 47.17 (12.05)
  MCS-WK72 (n=45) | 49.45 (10.26)
  MCS Change from BL (n=45) | 0.54 (11.51)

2. Primary Outcome: Change From Baseline (BL) to Week 72 (WK72) in Chronic Liver Disease Questionnaire-Hepatitis C Virus (CLDQ-HCV)
Description: The CLDQ-HCV is a disease-specific questionnaire measuring HRQL that contains 29 items divided into 4 domains: emotional function (9 items), worry (6 items), systemic symptoms (8 items) and activity/energy (6 items). All items refer to the previous 2 weeks and are rated on a 7 point Likert scale, with 1 corresponding to the maximum frequency ("all of the time") and 7 to the minimum ("none of the time"). Domain scores are the means of the items contained. A summary score is calculated by the mean of all domain scores (CLDQ-HCV Global). Higher scores indicate better health-related quality of life.
Time Frame: Baseline, Week 72
Population: All Evaluable Participants (participants who had met the evaluation and eligibility criteria and were included in the study) who had CLDQ-HCV data available at baseline and Week 72.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEG + RBV (Standard Clinical Practice)
Number analyzed (Participants) | 125
score on a scale
  Activity/Energy-BL (n=125) | 5.58 (1.33)
  Activity/Energy-WK72 (n=46) | 5.76 (1.11)
  Activity/Energy Change from BL (n=46) | -0.06 (1.16)
  Emotional Function-BL (n=125) | 5.19 (1.02)
  Emotional Function-WK72 (n=46) | 5.35 (0.97)
  Emotional Function Change from BL (n=46) | 0.10 (0.87)
  Worry-BL (n=125) | 5.26 (1.25)
  Worry-WK72 (n=46) | 5.65 (1.46)
  Worry Change from BL (n=46) | 0.41 (1.21)
  Systemic Symptoms-BL (n=125) | 5.25 (1.18)
  Systemic Symptoms-WK72 (n=46) | 5.57 (1.06)
  Systemic Symptoms Change from BL (n=46) | 0.09 (0.80)
  CLDQ-HCV Global -BL (n=125) | 5.31 (1.06)
  CLDQ-HCV Global-WK72 (n=46) | 5.56 (1.05)
  CLDQ-HCV Global Change from BL (n=46) | 0.15 (0.87)
Statistical Analysis 1: Comparison: PEG + RBV (Standard Clinical Practice); Within-group comparison of Worry domain between BL Visit and WK72 Visit; Test type: Superiority or Other; p = 0.027, Student´s t-test for paired samples

3. Secondary Outcome: Change From Baseline to Week 72 (WK72) in SF-36 Scores Among Participants Who Completed Treatment and Participants Who Had Early End of Treatment (Subset Analysis)
Description: as for outcome 1
Time Frame: Baseline, Week 72
Population: All Evaluable Participants (participants who had met the evaluation and eligibility criteria and were included in the study) who had SF-36 data available at baseline and Week 72. Analysis Population included 38 participants who completed 48 weeks of treatment and 8 participants who did not complete 48 weeks of treatment (early end).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PEG + RBV (Standard Clinical Practice): Completed Treatment: Participants who completed 48 weeks of PEG and RBV in combination therapy according to standard clinical practice followed by 24 weeks of observation.
- PEG + RBV (Standard Clinical Practice): Early End of Treatment: Participants who did not complete 48 weeks of PEG and RBV in combination therapy according to standard clinical practice but instead had an early end of treatment. Treatment was followed by 24 weeks of observation.
Arm/Group | PEG + RBV (Standard Clinical Practice): Completed Treatment | PEG + RBV (Standard Clinical Practice): Early End of Treatment
Number analyzed (Participants) | 38 | 8
score on a scale
  Physical Function (n=37, n=8) | -1.08 (17.88) | -3.75 (4.43)
  Physical Role (n=37, n=8) | -1.35 (38.62) | 3.13 (8.84)
  Pain (n=38, n=8) | -3.55 (19.32) | 4.13 (17.75)
  General Health (n=38, n=8) | 4.35 (19.38) | -10.00 (16.42)
  Vitality (n=37, n=8) | -1.98 (21.54) | -15.00 (19.09)
  Social Function (n=38, n=8) | 4.61 (22.40) | -9.38 (20.86)
  Emotional Role (n=37, n=8) | 4.50 (40.19) | -12.50 (35.36)
  Mental Health (n=37, n=8) | 3.46 (17.41) | -9.50 (25.38)
  PCS (n=37, n=8) | -1.23 (6.51) | 0.59 (5.90)
  MCS (n=37, n=8) | 2.18 (11.01) | -7.05 (11.36)
Statistical Analysis 1: Comparison: PEG + RBV (Standard Clinical Practice): Completed Treatment vs PEG + RBV (Standard Clinical Practice): Early End of Treatment; Between-group comparison of change from baseline in MCS; Test type: Superiority or Other; p = 0.038, Student´s t-test for paired samples

4. Secondary Outcome: Change From Baseline to Week 72 (WK72) in CLDQ-HCV Scores Among Participants Who Completed Treatment and Participants Who Had Early End of Treatment (Subset Analysis)
Description: The CLDQ-HCV is a disease-specific questionnaire measuring quality of life that contains 29 items divided into 4 domains: emotional function (9 items), worry (6 items), systemic symptoms (8 items) and activity/energy (6 items). All items refer to the previous 2 weeks and are rated on a 7 point Likert scale, with 1 corresponding to the maximum frequency ("all of the time") and 7 to the minimum ("none of the time"). Domain scores are the means of the items contained. A summary score is calculated by the mean of all domain scores (CLDQ-HCV Global). Higher scores indicate better health-related quality of life.
Time Frame: Baseline, Week 72
Population: All Evaluable Participants (participants who had met the evaluation and eligibility criteria and were included in the study) who had CLDQ-HCV data available at baseline and Week 72. Analysis Population included 38 participants who completed 48 weeks of treatment and 8 participants who did not complete 48 weeks of treatment (early end).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEG + RBV (Standard Clinical Practice): Completed Treatment | PEG + RBV (Standard Clinical Practice): Early End of Treatment
Number analyzed (Participants) | 38 | 8
score on a scale
  Activity/Energy (n=38, n=8) | 0.04 (1.17) | -0.50 (1.07)
  Emotional Function (n=38, n=8) | 0.25 (0.83) | -0.57 (0.72)
  Worry (n=38, n=8) | 0.61 (1.18) | -0.58 (0.82)
  Systemic Symptoms (n=38, n=8) | 0.15 (0.82) | -0.23 (0.58)
  CLDQ-HCV Global (n=38, n=8) | 0.28 (0.86) | -0.49 (0.67)
Statistical Analysis 1: Comparison: PEG + RBV (Standard Clinical Practice): Completed Treatment vs PEG + RBV (Standard Clinical Practice): Early End of Treatment; Between-group comparison of change from baseline in Emotional Function domain; Test type: Superiority or Other; p = 0.014, Student´s t-test for paired samples
Statistical Analysis 2: Comparison: PEG + RBV (Standard Clinical Practice): Completed Treatment vs PEG + RBV (Standard Clinical Practice): Early End of Treatment; Between-group comparison of change from baseline in Worry domain; Test type: Superiority or Other; p = 0.009, Student´s t-test for paired samples
Statistical Analysis 3: Comparison: PEG + RBV (Standard Clinical Practice): Completed Treatment vs PEG + RBV (Standard Clinical Practice): Early End of Treatment; Between-group comparison of change from baseline in CLDQ-HCV Global domain; Test type: Superiority or Other; p = 0.022, Student´s t-test for paired samples

5. Secondary Outcome: Minimal Clinically Important Difference (MCID) in SF-36 Scores
Description: SF-36 is a 36-item questionnaire measuring HRQL covering 2 summary measures, PCS and MCS. The SF-36 consists of 8 subscales. PCS is represented by physical function, role limitations-physical, pain, and general health perception. MCS is represented by vitality, social function, role limitations-emotional, and mental health. Subscale items are summed and scaled from 0-100 to give subscale scores; 0= worst HRQL, 100=best HRQL. PCS and MCS summary scores are constructed as T-scores (mean =50, standard deviation=10) with no minimum or maximum score; higher scores indicate better health status. MCID was defined as the difference in questionnaire scores between baseline and final visits for those participants who had stated that their health status had changed at the end of the study (improved in one category of health status as perceived by themselves). The MCID was calculated for each subscale of the SF-36 and for PCS and MCS.
Time Frame: From Baseline Visit to Final Visit (up to 72 weeks)
Population: All Evaluable Participants (participants who had met the evaluation and eligibility criteria and were included in the study) who had improved in one category of health status as perceived by themselves.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEG + RBV (Standard Clinical Practice)
Number analyzed (Participants) | 7
score on a scale
  Physical Function | 4.29 (16.44)
  Physical Role | 3.57 (50.89)
  Pain | -0.67 (39.00)
  General Health | 6.86 (13.31)
  Vitality | 4.29 (29.64)
  Social Function | -5.36 (17.47)
  Emotional Role | 14.29 (37.80)
  Mental Health | 4.57 (13.35)
  PCS | 0.19 (6.76)
  MCS | 2.73 (9.43)

6. Secondary Outcome: MCID in CLDQ-HCV Scores
Description: The CLDQ-HCV is a disease-specific questionnaire measuring HRQL that contains 29 items divided into 4 domains: emotional function (9 items), worry (6 items), systemic symptoms (8 items) and activity/energy (6 items). All items refer to the previous 2 weeks and are rated on a 7 point Likert scale, with 1 corresponding to the maximum frequency ("all of the time") and 7 to the minimum ("none of the time"). Domain scores are the means of the items contained. A summary score is calculated by the mean of all domain scores (CLDQ-HCV Global). Higher scores indicate better health-related quality of life. MCID was defined as the difference in questionnaire scores between baseline and final visits for those participants who had stated that their health status had changed at the end of the study (improved in one category of health status perceived by themselves). The MCID was calculated for each domain of the CLDQ-HCV and for the CLDQ-HCV summary score.
Time Frame: From Baseline Visit to Final Visit (up to 72 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEG + RBV (Standard Clinical Practice)
Number analyzed (Participants) | 7
score on a scale
  Activity/Energy | 0.00 (1.58)
  Emotional Function | 0.40 (0.64)
  Worry | 1.00 (0.84)
  Systemic Symptoms | 0.00 (0.71)
  CLDQ-HCV Global | 0.40 (0.83)

7. Secondary Outcome: Percentage of Participants Who Were Compliant With Treatment According To Medication Count (Subset Analysis)
Description: Compliance was calculated as the amount of dispensed medication minus the amount of medication returned by participants divided by amount of dispensed medication.
Time Frame: From Baseline Visit to Final Visit (up to 72 weeks)
Population: All Evaluable Participants; participants who had met the evaluation and eligibility criteria and were included in the study. Analysis Population included 53 participants who completed 48 weeks of treatment and 77 participants who did not complete 48 weeks of treatment (early end).
Measure: Number; unit: percentage of participants
Arm/Group | PEG + RBV (Standard Clinical Practice): Completed Treatment | PEG + RBV (Standard Clinical Practice): Early End of Treatment
Number analyzed (Participants) | 53 | 77
percentage of participants
  PEG | 98.1 (1.17) | 0 (1.07)
  RBV | 81.1 (0.83) | 0 (0.72)
  PEG + RBV | 81.1 (1.18) | 0 (0.82)

ADVERSE EVENTS:
Time Frame: From Baseline visit to Final Visit (up to 72 weeks)
Description: Of 133 enrolled participants, AEs were collected for the 130 evaluable participants. 3 enrolled participants who failed screening did not have AEs reported.
Arm/Group | PEG + RBV (Standard Clinical Practice)
Serious Adverse Events (participants affected / at risk) | 12/130
Other Adverse Events (participants affected / at risk) | 116/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG + RBV (Standard Clinical Practice) (N=130)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4)
APLASIA PURE RED CELL (Blood and lymphatic system disorders) | 1 (1)
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 (1)
LYMPHOCYTIC INFILTRATION (Blood and lymphatic system disorders) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG + RBV (Standard Clinical Practice) (N=130)
ANAEMIA (Blood and lymphatic system disorders) | 7 (14)
NAUSEA (Gastrointestinal disorders) | 45 (70)
ASTHENIA (General disorders) | 19 (25)
FATIGUE (General disorders) | 34 (63)
INJECTION SITE REACTION (General disorders) | 61 (116)
PYREXIA (General disorders) | 19 (22)
WEIGHT DECREASED (Investigations) | 76 (140)
DECREASED APPETITE (Metabolism and nutrition disorders) | 10 (10)
MYALGIA (Musculoskeletal and connective tissue disorders) | 76 (153)
HEADACHE (Nervous system disorders) | 74 (146)
DEPRESSION (Psychiatric disorders) | 7 (9)
EMOTIONAL DISORDER (Psychiatric disorders) | 16 (18)
INSOMNIA (Psychiatric disorders) | 16 (18)
MENTAL DISORDER (Psychiatric disorders) | 25 (35)
ALOPECIA (Skin and subcutaneous tissue disorders) | 44 (73)
DRY SKIN (Skin and subcutaneous tissue disorders) | 13 (14)
PRURITUS (Skin and subcutaneous tissue disorders) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study data/results may not be published or disseminated without prior consent from the study sponsor. All publications arising from the study will cite all the participating researchers.